CLINICAL TRIAL: NCT03880604
Title: Triple Tourniquets With or Without IV Tranexamic Acid for Reducing Blood Loss at Open Myomectomy: A Double-blinded Randomized Placebo-controlled Trial
Brief Title: Triple Tourniquets With or Without Tranexamic Acid for Reducing Blood Loss at Open Myomectomy
Acronym: TTT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Aswan University Hospital (Other)
Responsible Party: Principal Investigator, hany farouk, Principal Investigator, Aswan University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: aswu/207/19
Record Dates: First submitted 2019-03-15; First posted 2019-03-19 (Actual); Last update posted 2019-05-13 (Actual); Status verified 2019-05

CONDITIONS: Myoma
Keywords: Haemostatic tourniquets; tranexamic acid; myomectomy
MeSH Terms: conditions — Myoma

STUDY DESIGN:
Intervention Model Description: A double-blinded randomized placebo-controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: A double-blinded randomized placebo-controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Triple tourniquets plus TA (Active Comparator): A number 1 polyglactin suture was tied around the cervix to occlude the uterine arteries, and polythene tourniquets were tied around the infundibulopelvic ligament to obstruct the ovarian vessels.plus1-gram tranexamic acid (10 ml) in 100 ml saline infusion
  Interventions: Procedure: Triple tourniquets; Drug: TA
- Triple tourniquets plus placebo to TA (Active Comparator): A number 1 polyglactin suture was tied around the cervix to occlude the uterine arteries, and polythene tourniquets were tied around the infundibulopelvic ligament to obstruct the ovarian vessels.plus placebo to 1-gram tranexamic acid (10 ml) in 100 ml saline infusion
  Interventions: Procedure: Triple tourniquets; Other: placebo to TA

INTERVENTIONS:
Procedure: Triple tourniquets — A number 1 polyglactin suture was tied around the cervix to occlude the uterine arteries, and polythene tourniquets were tied around the infundibulopelvic ligament to obstruct the ovarian vessels
  Other Names: Active comparator
Drug: TA — 1-gram tranexamic acid (10 ml) in 100 ml saline infusion
  Other Names: Active Comparator
  Arms: Triple tourniquets plus TA
Other: placebo to TA — placebo to 1-gram tranexamic acid (10 ml) in 100 ml saline infusion
  Other Names: placebo comparator
  Arms: Triple tourniquets plus placebo to TA

SUMMARY:
In this study, the investigators will investigate the effectiveness of an intravenous tranexamic acid plus triple tourniquets compared with triple tourniquets alone for the reduction of blood loss at the time of myomectomy

DETAILED DESCRIPTION:
An RCT investigated the efficacy of intravenous tranexamic acid (TA) during abdominal myomectomy. The study was unable to demonstrate any significant impact on blood loss, duration of surgery or need for blood transfusionHemostatic tourniquets to reduce intra-operative bleeding have long been available, but data on their efficacy from controlled trials are lacking. The investigators set out to evaluate the use of triple tourniquets plus tranexamic acid in controlled conditions and for the first time to investigate the hypothesis that adding tranexamic acid to tourniquet around the uterine artery reduces postoperative bleeding from the uterine incisions, a well-recognized sequel to surgery

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting for abdominal myomectomy with documented uterine fibroids on ----pelvic imaging
* Age ≥ 18 years and ≤ 50 years
* Pre-operative hemoglobin >8 g/dl
* Ability to understand and the willingness to sign a written informed consent.
* Admissible medical/surgical history
* Five or less symptomatic uterine myomas
* All myomas are subserous or intramural.
* Uterine size less than 24 weeks of pregnancy

Exclusion Criteria:

* Patients who have had a prior abdominal myomectomy
* Post-menopausal women
* Patients with known bleeding/clotting disorders
* Patients with a history of gynecologic malignancy
* Hypertension.
* Cardiac and Pulmonary Diseases.
* Obesity (body mass index > 30 kg/m2).
* History of allergic reactions attributed to misoprostol
* Cases that will require intraoperative conversion of myomectomy to hysterectomy

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — All women who prepared for abdominal myomectomies will be invited to participate in the study
Enrollment: 100 (Estimated)
Dates: Start 2019-04-01 (Actual); Primary Completion 2021-03-30 (Estimated); Study Completion 2021-07-01 (Estimated)

PRIMARY OUTCOMES:
Mean amount of intraoperative blood loss | intraoperative
  measure the mean amount of intraoperative blood loss by gravimetric methods

SECONDARY OUTCOMES:
The number of patients needs for blood transfusion | 24 hours post delivery
  Calculation the number of patients needs for blood transfusion

CONTACTS AND LOCATIONS:
Overall Officials: hany f sallam, md, Principal Investigator — Aswan University Hospital
Locations (1):
- Aswan University Hospital, Aswān, Egypt

IPD SHARING:
Plan to Share IPD: No